CLINICAL TRIAL: NCT04891029
Title: Phase III Diagnostic Trial for Early Detection of Endometrial/Ovarian Cancer and Hereditary Predisposition of These Cancers
Brief Title: Early Detection of Endometrial/Ovarian Cancer and Hereditary Predisposition of These Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Genome Canada (Other); Genome Quebec (Other); Research Institute of the McGill University Health Center (Unknown); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Lucy Gilbert, Professor Department of Obstetrics & Gynecology and Department of Oncology, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-6430
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Diagnoses Disease
Keywords: Ovarian Cancer; Endometrial Cancer; Genomics; Screening; Early detection
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: DOvEEgene test — Women participating in the study will undergo a genomic uterine pap test, DOvEEgene test, for the screening of ovarian and endometrial cancers. Clinical tests will also be administered as a comparator (CA-125 blood test and TVUS).

SUMMARY:
Early stage high-grade cancer, endometrial and ovarian, has few, if any, symptoms or signs. When symptoms appear, the disease is commonly in advanced stage meaning it has left the gynaecological organs and metastasized to the pelvic/abdominal cavity. The McGill research group had showed in the DOvEE trial (NCT02296307), that fast-track assessment with transvaginal ultrasound scans (TVUS) and serial CA125 of women with vague symptoms associated with ovarian and endometrial cancer did diagnose these cancers earlier in the disease trajectory, with low-volume resectable disease, but only after the cancer had already become Stage III. One way to detect these cancers earlier is to screen asymptomatic women. Unfortunately, none of the currently available tests, including TVUS and CA-125 have been shown to be useful for screening for ovarian or endometrial cancer.

The McGill team has developed a genomic assay to screen and detect these cancers earlier in the trajectory than is currently the case. The test identifies pathogenic somatic mutations (necessary early steps in the development of these cancers), in an uterine cytological sample. It is able to do so by incorporating a machine-learning derived classifier that can discriminate the mutational signature of these cancers from benign disease with a sensitivity of 80% and a specificity of 100% in a healthy population of peri- and post-menopausal women. In addition to the uterine sample, the test includes a saliva sample that acts as an internal control but can also identify germline pathogenic variants that predispose to hereditary endometrial/ovarian cancers as well as breast, pancreas, and colon cancers.

The test was developed in a retrospective population in whom the assay was done pre-operatively and the diagnosis of malignancy versus benign gynecological disease was confirmed by detailed pathological analysis of the uterus, tubes, and ovaries after surgical resection (NCT02288676). The test is now ready to be tested as a phase III diagnostic test in the general population to see if these results are just as promising in the community at large.

ELIGIBILITY:
Inclusion Criteria:

- Capacity to understand study and provide informed consent

Exclusion Criteria:

* Prior hysterectomy
* Be pregnant
* Be nursing
* Be undergoing any fertility treatment
* Have had recent history of uterine perforation

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5600 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Early diagnosis of ovarian and endometrial cancers | 3 years
  Through the identification of pathogenic somatic mutations in uterine pap sample in combination with an established machine learning algorithm, the team will discriminate cancer from benign disease in participant samples.
Identification of germline mutations | 3 years
  To determine the proportion of the study population who are carriers of clinically significant pathogenic germline mutations.

SECONDARY OUTCOMES:
Evaluate women's experience related to study procedures | 3 years
  Assess women's experience to the genomic uterine pap sampling process using an acceptability questionnaire. It is important the participant has a good experience with the sampling and healthcare professional.
Evaluate effects on quality of life from study participation | 3 years
  We will assess effects on quality of life (QoL) to study participants, such as anxiety while awaiting results, interventions for false positives results and etc. via the SF-36 questionnaire.
Evaluate costs of unnecessary intervention | 3 years
  We will track the cost of every intervention resulting from a positive test, till we determine whether it was a false positive or not. For instances of a false positive result, we will consider the associated costs via a health economics analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - McGill University Health Centre, Royal Victoria Hospital, Montreal, Quebec
  - Queen Elizabeth Health Complex, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No